CLINICAL TRIAL: NCT03793803
Title: Clinical Trial of Home Palliative Care for Seriously Ill Adults
Brief Title: Trial of Mount Sinai Palliative Care at Home
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Nathan Goldstein, Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: GCO 15-2215
Record Dates: First submitted 2018-12-24; First posted 2019-01-04 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Organ Failure
Keywords: Palliative Care; Home-Based Care

STUDY DESIGN:
Intervention Model Description: Patients and caregivers are randomized to receive care from the home-based palliative care team or will receive usual care from their primary physician
Who Masked: Outcomes Assessor
Masking Description: Single Blind Control - Outcomes assessor is blind to randomization arms
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home Palliative Care (Experimental): Randomized to Intervention Arm
  Interventions: Behavioral: Home Palliative Care
- Control Arm (No Intervention): Usual Care - Patients will be cared for by the physician who treats their primary illness(es).

INTERVENTIONS:
Behavioral: Home Palliative Care — Patients/caregivers will be cared for by an interdisciplinary team that includes a social worker, nurse, community health worker, nurse practitioner, and physician.
  Arms: Home Palliative Care

SUMMARY:
The proposed project is a randomized controlled trial of a new home-based palliative care program for adults with serious illness and their caregivers within the Mount Sinai Health System. Potential subjects will be identified from Mount Sinai records or referred by a Mount Sinai healthcare provider. Patients will only be approached after authorization by their Mount Sinai physician. Participants who consent to enrollment will be randomized to receive the intervention (home-based palliative care program) or usual care (with their nominated Mount Sinai physician). Patients will be enrolled in the study for a minimum of 6 months.

After 6 months, patients can remain in the program if there is ongoing clinical need; data collection beyond 6 months will be done on all patients through chart abstraction/ administrative claims only.

Effectiveness of the intervention will be determined through assessment of patient and caregiver reported outcomes and abstraction of data from medical records and administrative claims. Impact on the following parameters will be measured: (i) Patient symptoms, quality of life, satisfaction with care, documentation of advanced directives, receipt of care consistent with preferences (ii) Caregiver burden, satisfaction with care, and depression (iii) Healthcare utilization and costs of care.

DETAILED DESCRIPTION:
The objective of this randomized controlled trial is to study the impact of a new home based palliative care program on patients' symptoms, quality of life, satisfaction with care, completion of advance care planning documentation and receipt of care consistent with preferences. In addition, the study will examine the impact of this model of care on patient healthcare utilization, including hospitalization, emergency department utilization, and hospice use prior to death. The trial will also include patients' caregivers, in order to examine the impact of the intervention on caregiver burden and prevalence of depression.

Patients randomized to the intervention will be scheduled for an intake visit. This visit will be undertaken by the team's registered nurse and/or social worker, together with a community health worker, and other team members (advanced practice nurse, MD), depending on patients' needs. Following this visit, and in conjunction with the nurse practitioner and/or MD, a care plan will be developed to address areas of clinical need highlighted during the intake visit.

Patients in the intervention arm will receive ongoing monitoring and input (telephone-based and in-person) from members of the clinical team, dependent on their identified needs. Patients' cases will be discussed at the weekly IDT meeting, as appropriate to the level of clinical need. Patients and caregivers will be provided with access to a 24 hour telephone line, staffed by a Mount Sinai based physician, which acts as an advice line out of hours. These physicians will be able to provide advice to patients and caregivers.

ELIGIBILITY:
Inclusion Criteria:

* Presence of a "serious medical illness" - according to pre-specified diagnostic code-based criteria
* Subject has a Mount Sinai physician who authorizes their participation in the study and receipt of the program
* Subject is resident in Manhattan outside of a long term care facility and is not receiving hospice 5.
* Subject has evidence of capacity to benefit from enrollment in palliative care program
* Subject is conversant in English or Spanish
* Subject has capacity to consent

Exclusion Criteria:

* Subject has no usual physician within Mount Sinai
* Subject's usual physician doesn't provide authorization to patient participation
* Subject resident outside of Manhattan or in long term care facility or receiving hospice
* Subject is not conversant in English or Spanish
* Subject cannot provide informed consent to participation
* Dementia (where the subject does not have the capacity to consent)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 193 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
Integrated Palliative Outcomes Scale | 6 months
  Patient symptoms determined by the Integrated Palliative Outcomes Scale, a validated structured questionnaire administered to patient-subjects via telephone interview or in person by the trained research coordinator. The Integrated Palliative Outcomes Scale is scored on a likert scale from 0-4, with higher score indicating worse symptoms.

SECONDARY OUTCOMES:
McGill quality of life-revised | 6 months
  McGill quality of life-revised is a 14 item instrument administered to patient-subjects via telephone interview or in person by the trained research coordinator. Each item score on likert scale from 0-10, full scale from 0-140 with higher score indicating better quality of life.
Family Satisfaction with End-of-Life Care (FAMCARE-10) | 6 months
  FAMCARE-10 to assess patient satisfaction by using a validated 10-item structured questionnaire administered to patient-subjects via telephone interview or in person by the trained research coordinator. FamCare each item score on likert scale 0-3, total scale from 0-30, with higher score indicating higher satisfaction
Number of Completion of Advance Directives | 6 months
  Study team will examine the patient's chart for completion of advanced directives.
Number of Preference Consistent Care | 6 months
  Study team will examine if the care patients receive is concordant with the care they wanted to receive. simple chart review of whether care received matches stated preferences (yes/no).
Zarit Burden Inventory | 6 months
  Zarit Burden Inventory to determine caregiver burden by using a validated structured 22-item questionnaire administered to caregiver-subjects via telephone interview or in person by the trained research coordinator. Each item is on a 5-point score range from 0 (never) to 4 (always). Full scale from 0 to 88, with higher score indicating more burden.
FAMCARE-10 | 6 months
  FAMCARE-10 to assess caregiver satisfaction by using a validated 10-item structured questionnaire administered to patient-subjects via telephone interview or in person by the trained research coordinator. FamCare each item score on likert scale 0-3, total scale from 0-30, with higher score indicating higher satisfaction.
The Patient Health Questionnaire (PHQ-9) | 6 months
  PHQ-9 to assess Caregiver Depression by using a validated structured 9 item questionnaire administered to caregiver-subjects via telephone interview or in person by the trained research coordinator. The PHQ-9 is the depression module, which scores each of the 9 DSM-IV criteria as "0" (not at all) to "3" (nearly every day). Full scale from 0-27, with higher score indicating worse depression.
Number of inpatient admissions | 6 months
  Number of inpatient admissions to measure healthcare utilization
Number of emergency department visits | 6 months
  Number of emergency department visits to measure healthcare utilization
Number of outpatient appointments | 6 months
  Number of outpatient appointments to measure healthcare utilization

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Goldstein, MD, Study Director — Icahn School of Medicine at Mount Sinai
Locations (4):
- United States (4):
  - Mount Sinai Beth Israel, New York, New York
  - Mount Sinai West, New York, New York
  - Mount Sinai St Luke's, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York

IPD SHARING:
Plan to Share IPD: No